CLINICAL TRIAL: NCT06814600
Title: Prevalence of Non-Alcoholic Fatty Liver Disease in Inflammatory Bowel Disease Patients: A Prospective Monocentric Study
Brief Title: Prevalence of Non-Alcoholic Fatty Liver Disease in Inflammatory Bowel Disease Patients
Acronym: PONI
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Jennifer Aoun, Medical doctor, Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: PONI
Record Dates: First submitted 2025-01-30; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: NAFLD; Inflammatory Bowel Diseases; Steatosis; Fibrosis, Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Inflammatory Bowel Diseases; Fatty Liver; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Baseline assessment: All patients with a confirmed diagnosis of IBD (cf. inclusion criteria) will have their demographic and clinical data collected during consultation via the medical record system Xcare/Abrumet. This include their age, gender, ethnicity, calculated BMI, alcohol consumption, smoking history, medical history (Hypertension, diabetes type II and dyslipidemia) and surgical history.
  Clinical data such as disease type, duration and IBD related current medications will be noted. The gastroenterologist will fill an assessment questionnaire in order to clinically assess the disease activity. This consists of Partial Mayo clinical score (pMayo) for Ulcerative Colitis and Harvey Bradshaw Index (HBI) for Crohn's disease. Remission is defined as a pMayo ≤ 1 or a HBI <5, mild disease is defined as pMayo between 2 and 4, or HBI between 5 and 7. Finally, moderate to severe disease is defined as pMayo ≥ 5, or HBI > 85.
  According to the data provided, patients will be classified into two sub-groups accor
  Interventions: Diagnostic Test: Transient elastometry
- Follow-up Assessment: Patients selected in the phase A of the study will be followed over time, through the course of their disease following the usual protocol for IBD patients follow up.
  They will undergo the same assessment when a change in the baseline intestinal disease activity occurs: This is defined as a progression from remission state to active disease state or vice versa.
  The assessment consists of the clinical questionnaire to be filled by the gastroenterologist during a follow up consultation (pMayo and HBI), routine blood tests for biochemical follow up of the disease activity, measurements of cytokines and inflammatory proteins (similar to phase A), FIB-4 score calculation and a repeat transient elastometry "Fibroscan".
  Interventions: Diagnostic Test: Transient elastometry

INTERVENTIONS:
Diagnostic Test: Transient elastometry — Controlled attenuation parameter (CAP) and liver stiffness measurement (LSM) will be measured by transient liver elastometry "Fibroscan" to evaluate hepatic steatosis and fibrosis in all patients at baseline. Absence of steatosis S0 is defined as CAP <248 dB/m, mild steatosis S1 with CAP < 268 dB/m, and moderate to severe steatosis ≥ S2 is defined as CAP >280 dB/m. Liver fibrosis will be evaluated using the liver stiffness measurement (LSM) in kPa7.

SUMMARY:
Non-alcoholic Fatty Liver Disease (NAFLD) refers to a spectrum of disease characterized by the presence of more than 5% of steatosis in hepatocytes of individuals who consume little or no alcohol. It ranges from simple steatosis without evidence of inflammation, to the association of steatosis and inflammation with cellular necrosis, the so-called non-alcoholic steatohepatitis (NASH). NAFLD has become increasingly common in developed countries affecting up to 38% of the population. It is mostly but not exclusively associated with metabolic syndrome including obesity, insulin resistance, and hypertension. There is growing evidence of a close interaction between the gut and the liver "Gut-liver axis", particularly in the pathogenesis of NAFLD. The pathophysiological mechanism behind this association is not well understood but involves small intestinal bacterial overgrowth (SIBO), intestinal wall inflammation and increased permeability, all leading to systemic translocation of microbial metabolites including endotoxins and pro-inflammatory markers called Pathogen Associated Molecular Pattern (PAMPs). Thus, the gut-liver interaction, mediated by cytokines and inflammatory proteins seem to be the cornerstone of this complex liver disease.

Recent studies underlined the increased prevalence of NAFLD in the Inflammatory Bowel Disease (IBD) population, accounting for almost 32% of hepatic extra-intestinal manifestations of the disease. Several hypotheses have been proposed to explain the pathophysiology behind this association, encompassing chronic intestinal wall inflammation, increased intestinal permeability and altered gut microbiota or dysbiosis. To our knowledge, no studies have been conducted so far to investigate the correlation between intestinal disease activity (IBD flare versus remission state) and NAFLD incidence and behavior (progression versus regression of steato-fibrosis). We therefore aim to conduct a prospective paired study, on IBD patients followed at Saint-Pierre University Hospital, aiming to explore this correlation.

In this paired study design, patients will be their own controls over the course of their disease: An evaluation of NAFLD will be done for all patients during both phases of their inflammatory bowel disease: In the active phase and in remission phase. Our primary outcome is to assess NAFLD prevalence in the IBD population followed at our institution. Secondary outcomes will be to explore NAFLD prevalence and behavior (progression versus regression of steato-fibrosis) according to IBD activity, IBD type, IBD duration and types of IBD treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBD based on clinical, endoscopic, and histological gounds according to the latest ECCO guidelines
* Willingness to provide informed consent for study participation

Exclusion Criteria:

* Presence of established liver disease (including autoimmune hepatitis, primary biliary cholangitis, primary biliary cirrhosis, hemochromatosis, Wilson's disease, positive serology for viral hepatitis B or C)
* History of hepatocellular carcinoma or liver transplantation
* History of excessive alcohol consumption defined as >3 units per day for women and > 5 units per day for men
* Pregnancy at the time of recruitment
* Failure to perform an elastography mesure or missing elastography data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBD patients followed at Saint-Pierre University Medical Center, Brussels, Belgium
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NAFLD in the population of IBD patients followed at the University Hospital IBD clinic. | From enrollement to the end of the study, up to 12 months
  Prevalence of NAFLD in the population of IBD patients followed at the University Hospital IBD clinic.

SECONDARY OUTCOMES:
Behavior of NAFLD according to the IBD activity | From enrollement to the end of the study, up to 12 months
  Behavior of NAFLD (progression versus regression of steato-fibrosis) according to IBD activity (active disease versus remission)
NAFLD predictors in IBD patients | From enrollement to the end of the study, up to 12 months
  Independent predictors (risk factors) for NAFLD in our IBD patients study population such as particular demographics, IBD disease type, IBD disease duration, IBD treatments, patients' immunological profiles, and various inflammatory markers.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Saint Pierre, Brussels, Belgium